CLINICAL TRIAL: NCT01457079
Title: Keloid Radiation Registry
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Tirgan, Michael H., M.D. (Individual)
Responsible Party: Sponsor
Other Study IDs: Tirgan 11-06
Record Dates: First submitted 2011-10-19; First posted 2011-10-21 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-10

CONDITIONS: Keloid
Keywords: Keloid; Radiation Therapy; Hypertrophic Scar
MeSH Terms: conditions — Keloid; Cicatrix, Hypertrophic

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

SUMMARY:
Radiation therapy has been, and is being used in treatment of patients with keloid. Radiation is typically used as an adjunct to surgery in order to reduce the recurrence rate of keloid.

Radiation therapy is not free of long term side effects. Radiation Therapy is known to cause secondary cancers. The investigators also do not have a good understanding as to how effective radiation therapy is in preventing recurrence of keloid.

Purposes of this study are to determine the long term safety as well as efficacy of radiation therapy when used for treatment of keloid.

DETAILED DESCRIPTION:
The Keloid-Radiation project is a clinical registry of patients with keloid who have been treated with Radiation Therapy. This registry aims to monitor the at least 1,000 keloid patients who received radiation therapy to their keloid and to collect epidemiological and clinical data about these patients in order to assess the long term safety and effectiveness of radiation therapy.

Radiation is currently being used in the treatment of keloid, thus enabling the epidemiological characteristics of patients, analysis of treatment response, modeling the influence of risk factors on patients´ risk of developing long term complications such as a cancer, as well as the detailed analysis of the dose delivered, equipment used and radiation planning. This study intends to gather data about the long term efficacy and safety of radiation therapy and rate of developing secondary cancers in patients who have received radiation therapy for treatment of their keloid.

ELIGIBILITY:
Inclusion Criteria:

1. Clinically confirmed diagnosis of keloid
2. History of radiation therapy for treatment of keloid
3. All Ages
4. Signed informed consent form ( by parent or legal guardian if patient is under the age of 18)

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study intends to enroll all patients who have had, or will be receiving radiation therapy for their keloid(s).
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2011-12; Primary Completion 2020-12 (Estimated); Study Completion 2021-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Michael H Tirgan, MD, Study Chair — St. Luke's-Roosevelt Hospital Center
Locations (1):
- Michael H. Tirgan, MD, New York, New York, United States